CLINICAL TRIAL: NCT07178860
Title: Respiratory Health and Wellbeing Post Pulmonary Tuberculosis
Acronym: RESPOST
Status: Recruiting | Type: Observational
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 25009
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis (TB)
Keywords: Post-TB; TB; Tuberculosis; Post-tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We know that in low-income countries where there is a lot of tuberculosis (TB) about 20%-50% of people treated for TB have long term problems with their lungs and general wellbeing. This means they can't always get back to doing activities they were doing before they had TB and may need further treatment, for example antibiotics, inhalers or special rehabilitation classes. Some people are unnecessarily treated again for TB because they still have a cough. There have been two international guides published recently, describing standards for providing follow up care for people treated for TB. However, in the UK despite there being 4000 new cases of TB diagnosed every year, we do not follow these guidelines and we do not know if people treated for TB here have similar residual problems with their lungs and general wellbeing. It is difficult to advocate for people treated for TB to have follow up care if we do not know the size of the problem. Anecdotally, experts who do the clinics report that there are a large percentage of people who go on to have long term health problems after they are "cured" from TB but there is no pathway to follow them up. There are no UK guidelines or funding to support TB follow-up or ongoing treatment. It is possible, extrapolating from the data from other countries, that 2000 people a year in UK have undiagnosed or untreated lung health problems because of their previous TB.

We would like to see if people who are treated in the Liverpool TB service (a regional referral service) have long term problems with their lungs. We will do this by inviting people who were treated for TB to come for a review at approximately 1 year after finishing their treatment.

We will ask them to blow into a lung function testing machine (the same that is used for diagnosing asthma) and ask them questions about their health and wellbeing. If they have cough, we will ask them for a sputum sample, and we will collect a blood sample if people are willing to donate a small amount of blood to be used in future research. These will be stored in a special freezer for future related studies into biomarkers and mechanisms of disease.

We will also invite some people to partake in recorded interviews where they can give their opinion about how they feel having been treated for TB and what (if any) follow up they feel they would benefit from.

We hope that by recording the problems (if any) the people treated for TB have, we will then be able to use this data to design a larger UK-wide study investigating the prevalence of lung disease after treatment for TB. If we find that there is significant disease, in future we can then test treatment options and care pathways, as well as advocate for people to have improved follow up rather than just living with chronic lung health issues that might impair how well they can live their lives.

DETAILED DESCRIPTION:
There are over 10 million new diagnoses of tuberculosis (TB) annually and approximately 155 million TB survivors worldwide(1, 2). TB treatment varies but normally consists of 6 months of antimicrobial treatment, at the end of which the person is normally considered "cured" and discharged from the service. However, there is a growing body of evidence - including work led by study investigator (RN) - that suggests a significant number of survivors have morbidity that extends for years beyond TB treatment completion despite a "successful" treatment outcome(3-5). Approximately, half of individuals treated for pulmonary TB have some form of persistent pulmonary morbidity, with approximately 20% having significantly abnormal lung function(4, 5). Neurological, cardiac, psychological, and socioeconomic sequelae are also well recognised (6, 7). Following the 1st international symposium of Post-TB in Stellenbosch South Africa, in 2019, TB survivors called for researchers and clinicians to develop guidance and pathways for follow-up after TB treatment completion(8). In April 2023, a consortium of international experts published the first clinical statement on post-TB Health and Wellbeing(7). In addition, the minimum clinical standards for post-TB lung disease were published by the International Journal of Tuberculosis and Lung Disease, highlighting the need for ongoing follow-up for survivors of tuberculosis(9).

The vast majority of the epidemiological and clinical data on post-TB lung disease comes from low- and middle-income countries with a high burden of TB, it is this data which has provided evidence for the new international clinical standards of care(7, 9).

The UK is a high-income country with low TB incidence compared to countries such as South Africa. However the burden of disease is not insignificant with over 4000 new diagnoses made annually(10). TB disproportionately affects vulnerable and disadvantaged populations and many affected have comorbidities which may increase the risk of ongoing PTLD(10, 11). The North-West region of England has seen a recent sharp rise in TB diagnoses, increasing by 11% in quarter 3 in 2023 compared to the same quarter in 2022(10). Despite this there is no published data on the burden of post-TB lung disease in the UK, and it is unknown if there are similarly high numbers of survivors with ongoing and untreated pulmonary symptoms. In the UK, the NICE guidelines for TB currently make no recommendation for follow-up care or treatment for Post-TB lung disease. There is potential for a large cohort of survivors with ongoing chronic lung disease but without a pathway to care in the UK. To advocate for the new clinical standards to become part of policy, the burden of disease first needs to be known.

Patient Participant Involvement (PPI) A patient expert, Fatima Karmadwala, who has survived drug-resistant TB, is a co-investigator. She has reviewed the information leaflet, consent form, lay summary and qualitative interview guides. She will attend study meetings and guide the team. This study idea originated from individuals who has survived TB and anecdotally told us they had ongoing symptoms here in the UK.

Rationale and Hypothesis There is an undescribed burden of post-TB lung disease in the UK that is similar to that seen in high-TB burden countries.

Rationale This is a pilot cross-sectional study that will allow us to describe the burden of post-TB lung disease in a population of TB survivors in Liverpool, UK. This data can then be used to design and accurately power a larger UK-wide epidemiological study, and if required implement a care pathway based on the already published international standards(7, 9).

Objectives

Primary objective:

1. To describe the prevalence of abnormal lung function in survivors of pulmonary-TB, 1 year after TB treatment completion.

   Secondary Objectives
2. To describe the prevalence of respiratory symptoms in survivors of pulmonary-TB, 1 year after TB treatment completion.
3. To describe the wider cost burden to TB survivors and their family (Adapted WHO TB patient cost survey).
4. To explore TB survivors' perspectives on the need for follow-up care for post-TB in Liverpool.
5. To support future pathogenesis and biomarker studies.

Study design Summary This is a cross-sectional observational design, focusing on adults, 18 years and older, who have been treated for pulmonary TB as part of the Liverpool regional TB service. After consent, participants will be asked to complete pre- and post-bronchodilator spirometry, demographic and symptoms questionnaire, a 6 minute walk test, the adapted WHO patient cost survey and subgroup will be asked if they would like to complete qualitative semi-structured interviews. Participants who have a productive cough will be asked to provide a sputum sample for mycobacterial investigation and storage. Participants willing to provide a blood sample will have blood collected. Ethical approval will be obtained from IRAS.

Study setting This is a single centre study carried out at Liverpool School of Tropical Medicine with recruitment from the Liverpool regional TB service which is based at the Liverpool University Hospitals NHS Foundation Trust. (Please note LSTM/LUHFT is a referral centre for the North-West and in some cases nationally for complex infectious disease cases including TB).

Study population A group of adults (over 18 years) who have completed treatment for pulmonary TB.

Inclusion Criteria:

1. Adults (over 18 years old)
2. Able to provide written informed consent
3. Previous diagnosis of microbiologically confirmed pulmonary TB
4. Completed TB treatment less than or equal to 18 months ago

Exclusion Criteria:

1. Previously diagnosed clinically significant chronic lung disease that is not well-controlled (for example COPD on significant treatment, or poorly controlled asthma)
2. Unable to perform spirometry due to contraindications to spirometry
3. Under the age of 18 years at the time of recruitment (not the time of initial diagnosis)
4. Incomplete history of TB treatment

Study procedures Identification and recruitment of participants Participants will be identified from Liverpool TB clinics, including the Liverpool TB Multidisciplinary Team (MDT) service that is co-chaired by co-investigators, Naomi Walker and Tom Wingfield. Participants will be approached in clinic at the end of their TB treatment or contacted via clinic letter or via their phone if that is their preferred method of communication. They will be invited to a research follow up clinic that is not part of their normal care. Posters will also be displayed in the TB-clinic and all clinic staff will be informed of the study and trained on the recruitment protocol. All potential participants will be given a participant information leaflet (PIL) and as much time as they need to consider it up until 18 months after TB treatment completion. All staff screening participants for eligibility will have had access to the patient records as part of the standard clinic work. Individuals will not be contacted about the study by staff who are not normally part of the TB clinic service until the point in which they have expressed an interest or agreed to being approached about the study by the clinical team. If the individual does not wish to take part, it will not affect their normal standard of care or have any effect on their TB treatment.

Screening for eligibility and enrolment At the time of obtaining consent

1. Participants will be asked questions to ensure they meet the inclusion criteria and do not meet any of the exclusion criteria: this may involve discussion about ongoing medical issues.
2. Where appropriate participants' medical notes will be reviewed by the study team to confirm that they meet the defined inclusion criteria.
3. The assessment of eligibility will be conducted by one of the research team who are formally delegated to do so by the Chief Investigator, are trained in GCP and understand the study protocol. Any queries about possible eligibility will be discussed with the Chief/Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* 1) Adults (over 18 years old) 2) Able to provide written informed consent 3) Previous diagnosis of microbiologically confirmed pulmonary TB 4) Completed TB treatment less than or equal to 18 months ago

Exclusion Criteria:

* 1) Previously diagnosed clinically significant chronic lung disease that is not well-controlled (for example COPD on significant treatment, or poorly controlled asthma) 2) Unable to perform spirometry due to contraindications to spirometry 3) Under the age of 18 years at the time of recruitment (not the time of initial diagnosis) 4) Incomplete history of TB treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult who have completed treatment for Pulmonary TB
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Abnormal Fev1 | Approximately 12 month Post TB treatment completion
  To describe the prevalence of abnormal lung function in survivors of pulmonary-TB, 1 year after TB treatment completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool School of Tropical Medicine, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data maybe sure fully anonymised for scientific reasons.
Supporting Information: Study Protocol